CLINICAL TRIAL: NCT02680808
Title: An Open Label Study in Healthy Volunteers to Evaluate the Potential for Cytochrome P450 3A4 Inhibition by F901318 Using Oral Midazolam as a Probe
Brief Title: Evaluation of the Potential for Cytochrome P450 3A4 Inhibition by F901318 Using Oral Midazolam as a Probe
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: F2G Biotech GmbH (Industry)
Collaborators: Hammersmith Medicines Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F901318.01.04.15
Record Dates: First submitted 2016-01-28; First posted 2016-02-12 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Invasive Aspergillosis
MeSH Terms: interventions — Midazolam; olorofim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- midazolam with F901318 (Experimental): Pharmacokinetic profile of midazolam 2 mg orally when given after dosing with F901318 to steady state.
  Interventions: Drug: Midazolam with F901318

INTERVENTIONS:
Drug: Midazolam with F901318 — Pharmacokinetics of midazolam with F901318

SUMMARY:
Open label evaluation of potential interaction of F901318 with cytochrome P450 3A4 using midazolam as a probe. Twenty healthy male subjects will participate

DETAILED DESCRIPTION:
This will be an open label study of midazolam (dose 2 mg orally, Day 1) followed by midazolam (2 mg orally) given after dosing with intravenous F901318 4 mg/kg bid for one day followed by 2.5 mg/kg bid for 7 doses (Day 7). Up to twenty subjects will be included in two cohorts which will undergo the same dosing schedules of midazolam and F901318 and undergo the same procedures. The first cohort will consist of 12 subjects studied in two groups of six subjects each. If there is clearly a difference in midazolam kinetics detectable between the first and second doses of midazolam, in this first cohort, the second cohort will not be studied. If there is no clear difference, the second cohort will also be studied to give a final result. PK sampling for midazolam and 1- and 4-hydroxymidazolam plasma and urine concentrations will continue for up to and including 24 hours after dosing with midazolam on both occasions. PK sampling for F901318 will continue from before the first dose and up to 24 hours after the ninth dose. A follow up visit will be conducted 7 +/- 2 days after discharge from the clinical unit following completion of blood sampling following the second dose of midazolam and the ninth dose of F901318.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will be males of any ethnic origin between 18 and 45 years of age and weighing 60-100 kg inclusive.
2. Subjects must be in good health, as determined by a medical history, physical examination, 12-lead electrocardiogram (ECG) and clinical laboratory evaluations (congenital non haemolytic hyperbilirubinaemia is acceptable).
3. Subjects will have given their written informed consent to participate in the study and to abide by the study restrictions.
4. Subjects must have ophthalmology assessments within the normal limits at screening. This includes normal Meibomian gland function.

Exclusion Criteria:

1. Male subjects who are not willing to use appropriate contraception during the study and for three months thereafter.
2. Subjects who have received any prescribed systemic or topical medication within 14 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
3. Subjects who have used any non-prescribed systemic or topical medication (including herbal remedies) within 7 days of the dose administration (with the exception of vitamin/mineral supplements and paracetamol) unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety.
4. Subjects who have received any medications, including St John's Wort, known to chronically alter drug absorption or elimination processes within 30 days of the dose administration unless in the opinion of the Investigator and the Medical Monitor the medication will not interfere with the study procedures or compromise safety. For at least 2 weeks prior to dosing and until all blood samples and observations are completed on Day 15 +/- 2s, subjects will not be allowed to eat any food or drink any beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family e.g. kale, broccoli, watercress, spring greens, kohlrabi, Brussels sprouts, mustard and charbroiled meats.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
area under concentration/time curve | 24 hours
  AUC0-24

SECONDARY OUTCOMES:
safety and tolerability as assessed by number of treatment related adverse events | 24 hours
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: FRANS VANDENBERG, Principal Investigator — Hammersmith Medicines Research
Locations (1):
- Hammersmith Medicines Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided